CLINICAL TRIAL: NCT03602586
Title: A Phase II Study of MK-3475 (Pembrolizumab) (NSC #776864) + Epacadostat (NSC #766086) in Recurrent Clear Cell Carcinoma of the Ovary
Brief Title: Testing Whether the Combination of Two Immunotherapy Drugs Have Activity in Recurrent or Persistent Clear Cell Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-01561; NCI-2018-01561 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY016 (Other: NRG Oncology); NRG-GY016 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2018-07-26; First posted 2018-07-27 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-06

CONDITIONS: Malignant Ovarian Clear Cell Tumor; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — epacadostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (epacadostat, pembrolizumab) (Experimental): Patients receive epacadostat PO BID and pembrolizumab IV over 30 minutes Q3W. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Epacadostat; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Epacadostat — Given PO
  Other Names: INCB 024360; INCB024360
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; QL2107; SCH 900475; SCH-900475; SCH900475

SUMMARY:
This phase II trial studies how well pembrolizumab and epacadostat work in treating patients with ovarian clear cell carcinoma that has come back (recurrent), remains despite treatment (persistent), or is growing, spreading, or getting worse (progressive). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Epacadostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab and epacadostat may work better compared to usual treatment (surgery, radiation, or cytotoxic chemotherapy) in treating patients with ovarian clear cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the objective tumor response (proportion of objective response by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) of the combination of pembrolizumab (MK-3475 [pembrolizumab]) and epacadostat in patients with recurrent or persistent clear cell carcinoma of the ovary.

SECONDARY OBJECTIVES:

I. To determine the nature and degree of toxicity of MK-3475 (pembrolizumab) + epacadostat as assessed by Common Terminology Criteria for Adverse Events (CTCAE) in patients with recurrent or persistent clear cell carcinoma of the ovary.

II. To estimate the progression-free survival (PFS) and overall survival (OS) in patients treated with combination of MK-3475 (pembrolizumab) and epacadostat.

EXPLORATORY TRANSLATIONAL OBJECTIVES:

I. Determine whether the ratio of plasma tryptophan to kynurenine (T:K) correlates with response to MK-3475 (pembrolizumab) + epacadostat, by evaluating plasma T:K pre-treatment, during treatment, and at disease progression.

II. Determine whether the presence of PD-L1, IDO-1, tumor-infiltrating regulatory T cells (Tregs), CD8 tumor-infiltrating lymphocytes (TILs), and human leukocyte antigen (HLA) class I in the tumor microenvironment at baseline correlates with objective response to MK-3475 (pembrolizumab) + epacadostat.

III. Determine whether soluble PD-L1 (sPD-L1) levels in plasma are correlated with response to MK-3475 (pembrolizumab) + epacadostat, by evaluating sPD-L1 concentrations pre-treatment, during treatment, and at disease progression.

OUTLINE:

Patients receive epacadostat orally (PO) twice daily (BID) and pembrolizumab intravenously (IV) over 30 minutes once every 3 weeks (Q3W). Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for 3 years, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Primary tumors must be at least 50% clear cell histomorphology in order to be eligible or have a histologically documented recurrence with at least 50% clear cell histomorphology. Recurrence should be biopsy proven as per standard of care unless the tumor is located in an area deemed unsafe to biopsy. Histologic confirmation of the original primary tumor is required via the pathology report. The percentage of clear cell histomorphology must be documented in the pathology report or in an addendum to the original report. If slides of the primary tumor are not available for review due to disposal of slides by the histology laboratory (typically 10 years after diagnosis), a biopsy of the recurrent or persistent tumor is required to confirm at least 50% clear cell histomorphology, as long as tumor is located in an area deemed safe to biopsy. The percentage of clear cell involvement must be documented in the pathology report or in an addendum to the original report
* All patents must have measurable disease, and at least one "target lesion" to be used to assess response as defined by RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray. Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 28 days prior to registration
  * Imaging of target lesions within 28 days prior to registration
  * Further protocol-specific assessments

    * Recovery from adverse effects of recent surgery, radiotherapy or chemotherapy (residual grade 1 toxicity is considered recovered)
    * Any other prior therapy directed at the malignant tumor including chemotherapy, and biologic/targeted agents must be discontinued at least 4 weeks prior to registration. Any hormonal therapy directed at the malignant tumor must be discontinued at least 2 weeks prior to registration
    * Any prior radiation therapy must be completed at least 4 weeks prior to registration, and progression must be outside the radiation field
    * At least 4 weeks must have elapsed since any major surgery prior to registration
* The trial is open only to women with recurrent or progressive clear cell carcinoma of the ovary
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 28 days prior to registration
* Patients must have had one prior platinum-based chemotherapy for management of primary disease. Patients are allowed to receive, but are not required to receive, up to two additional cytotoxic regimens for management of recurrent or persistent disease
* Absolute neutrophil count (ANC) >= 1,500/ul (within 14 days prior to registration)
* Platelets >= 100,000/ul (within 14 days prior to registration)
* Hemoglobin (Hgb) >= 8.0 g/dL within 14 days prior to registration (Note: the use of transfusion of other intervention to achieve a Hgb >= 8.0 g/dL is acceptable)
* Creatinine =< 1.5 x institutional upper limit of normal (ULN) or creatinine clearance (CrCl) >= 60 mL/min using Cockcroft-Gault formula (within 14 days prior to registration)
* Bilirubin =< 2.5 x ULN (within 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (within 14 days prior to registration)
* Normal thyroid function testing (thyroid-stimulating hormone [TSH]) (within 14 days prior to registration)
* Negative pregnancy test in women of childbearing potential
* Women of childbearing potential who are sexually active should be willing and able to use medically acceptable forms of contraception for the course of the study through 120 days after the last dose of MK-3475 (pembrolizumab). Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile, who have had a hysterectomy and/or bilateral oophorectomy) do not require contraception
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Patients who have had prior therapy with MK-3475 (pembrolizumab) or epacadostat or with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune check point pathways
* History of severe hypersensitivity reaction to any monoclonal antibody
* Patients with active auto-immune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease, Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure and unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures which are not controlled with non-enzyme inducing anticonvulsants, and/or epidural disease, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months prior to the first date of study treatment. Those with brain metastases are permitted as long as they have been treated with brain radiation therapy and have been documented stability 4 weeks following completion of brain radiation therapy
* In order for patients with human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) to be eligible, they must be on a stable highly active antiretroviral therapy (HAART) regimen with no drug-drug interaction with UGT1A9, have CD4+ counts > 350, with no detectable viral load on quantitative polymerase chain reaction (PCR), and no opportunistic infection
* Patients with treated hepatitis viral infections (hepatitis B and C) are eligible if they have completed definitive treatment at least 6 months prior, have no detectable viral load on quantitative PCR, and liver function tests (LFTs) meet eligibility requirements
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration
* Therapy with monoamine oxidase inhibitors (MAOIs) and selective serotonin reuptake inhibitor (SSRIs) within the last 4 weeks or history of serotonin syndrome. Concomitant use of monoamine oxidase inhibitors or SSRIs with epacadostat (INCB024360) is prohibited
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, abdominal/pelvic fistula, gastrointestinal perforation, gastrointestinal (GI) obstruction and/or who require parenteral hydration and/or nutrition
* Epacadostat (INCB024360) is a substrate of CYP3A4, CYP1A2, CYP2C19, UGT1A9, P-gp, and BCRP. Use caution when administered with strong inhibitors/inducers of these isoenzymes and transporter proteins. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference
* History or presence of an abnormal electrocardiography (ECG) that, in the investigator's opinion, is clinically meaningful. Screening QTc interval > 480 milliseconds is excluded (corrected by Fridericia). In the event that a single QTc is > 480 milliseconds, the subject may enroll if the average QTc for the 3 ECGs is < 480 milliseconds. For subjects with an intraventricular conduction delay (QRS interval > 120 msec), the JTc interval may be used in place of the QTc with sponsor approval. The JTc must be < 340 milliseconds if JTc is used in place of QTc. Subjects with left bundle branch block are excluded
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2024-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilian T Gien, Principal Investigator — NRG Oncology
Locations (363):
- United States (351):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - HaysMed, Hays, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Dickstein Cancer Treatment Center, White Plains, New York
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Puerto Rico (12):
  - Advance Oncology Center, Aguadilla
  - Doctor's Cancer Center-Arecibo, Arecibo
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Hematologia Oncologia San Pablo, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Primary Care Physician Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan
  - Centro de Hematologia y Oncologia del Sur, Santa Isabel

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Epacadostat, Pembrolizumab): Patients receive epacadostat PO BID and pembrolizumab IV over 30 minutes Q3W. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Epacadostat: Given PO (100 mg orally twice a day)
  Pembrolizumab: Given IV (200 mg IV infusion over 30 minutes Q3W)
Period: Overall Study
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Started | 14
Completed | 11
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete or Partial Objective Tumor Response
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v.) 1.1 criteria. Exact 95% confidence limits, accounting for interim analysis, will be provided in the final report. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=20% decrease in the sum of the longest diameter of target lesions and a 5 mm absolute increase; Overall Response (OR) = CR + PR.
Time Frame: Within 7 months of study entry
Population: Evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 14
Participants | 3

2. Secondary Outcome: Number of Participants With Adverse Events of Grade 3 or Higher
Description: Assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5. Number of participants with an adverse event of grade 3 or higher.
Time Frame: Adverse events were assessed from the start of treatment until 30 days after the end of the last treatment cycle. Adverse events were collected for a median time of 5.1 months and a maximum time of 23.8 months.
Population: All enrolled patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 14
Participants | 9

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Disease progression will be defined using RECIST v. 1.1 criteria. The distributions of PFS will be estimated and graphed using the Kaplan-Meier product limit method. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=20% decrease in the sum of the longest diameter of target lesions and a 5 mm absolute increase; Overall Response (OR) = CR + PR." Progression-free survival (PFS) is defined as the duration of time from the start of study treatment to time of progression or death, whichever occurs first.
Time Frame: Radiographic tumor assessments were completed 12 weeks after the start of treatment, then every 6 weeks for 49 weeks, followed by every 12 weeks until disease progression or treatment discontinuation. The median follow-up time was 4.8 months.
Population: Evaluable patients.
Measure: Number; unit: Participants with progression or death.
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 14
Participants with progression or death. | 14

4. Secondary Outcome: Overall Survival (OS)
Description: Assessment of deaths starting from the time of enrollment.
Time Frame: Overall survival (OS) is defined as the duration of time from the start of study treatment to time of death or the date of last contact. The median follow-up time for OS was 34.9 months.
Population: Evaluable patients.
Measure: Number; unit: Patients who died.
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 14
Patients who died. | 9

5. Other Pre Specified Outcome: Ratio of Plasma Tryptophan to Kynurenine (T:K)
Description: Will determine whether the ratio of plasma T:K correlates with response to MK-3475 (pembrolizumab) and epacadostat, by evaluating plasma T:K pre-treatment, during treatment, and at disease progression. Pre-treatment levels of T:K ratio in plasma will be assessed for association with radiographic response to MK-3475 (pembrolizumab) and epacadostat. Changes between pre-treatment and post-cycle 1 and changes between post-cycle 1 and disease progression for T:K ratio will be evaluated with paired Student's T tests.
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Presence of PD-L1, IDO-1, Tumor-infiltrating Regulatory T Cells (Tregs), CD8 Tumor-infiltrating Lymphocytes (TILs), and Human Leukocyte Antigen (HLA) Class I in the Tumor Microenvironment
Description: Will determine whether the presence of PD-L1, IDO-1, Tregs, CD8 TILs, and HLA class I in the tumor microenvironment at baseline correlates with objective response to MK-3475 (pembrolizumab) + epacadostat. Baseline presence of PD-L1, IDO-1, Tregs, TILs, and HLA class I in the tumor microenvironment will also be assessed for correlation with radiographic response to MK-3475 (pembrolizumab) and epacadostat. Will consider logistic regression models for these analyses of continuous biomarkers, if appropriate given the number of responses and if exact tests of response for categorized levels of the biomarkers.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Soluble PD-L1 (sPD-L1) Levels in Plasma
Description: Will determine whether sPD-L1 levels in plasma are correlated with response to MK-3475 (pembrolizumab) + epacadostat, by evaluating sPD-L1 concentrations pre-treatment, during treatment, and at disease progression. Pre-treatment levels of sPD-L1 in plasma will be assessed for association with radiographic response to MK-3475 (pembrolizumab) and epacadostat. Changes between pre-treatment and post-cycle 1 and changes between post-cycle 1 and disease progression for sPD-L1 will be evaluated with paired Student's T tests.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the start of treatment until 30 days after the end of the last treatment cycle. Adverse events were assessed from the start of treatment until 30 days after the end of the last treatment cycle. Adverse events were collected for a median time of 5.1 months and a maximum time of 23.8 months. All-Cause mortality was monitored/assessed for a longer time period than Adverse events. All-Cause Mortality monitored/assessed for a median of 34.9 months.
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 9/14
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Epacadostat, Pembrolizumab) (N=14)
Anemia (Blood and lymphatic system disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1
Ileal Obstruction (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Death Nos (General disorders) | 2
Inr Increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Ataxia (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Epacadostat, Pembrolizumab) (N=14)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 7
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 4
Blurred Vision (Eye disorders) | 1
Watering Eyes (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dry Mouth (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 8
Colitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Bloating (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Mucositis Oral (Gastrointestinal disorders) | 2
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Ileal Obstruction (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 4
Pain (General disorders) | 2
Malaise (General disorders) | 1
Flu Like Symptoms (General disorders) | 1
Fever (General disorders) | 3
General Disorders And Administration Site Conditio (General disorders) | 1
Fatigue (General disorders) | 11
Edema Limbs (General disorders) | 3
Death Nos (General disorders) | 2
Chills (General disorders) | 2
Allergic Reaction (Immune system disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Thrush (Infections and infestations) | 2
Vaginal Infection (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Shingles (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Bronchial Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Thyroid Stimulating Hormone Increased (Investigations) | 1
Platelet Count Decreased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 1
Inr Increased (Investigations) | 2
Creatinine Increased (Investigations) | 3
Cholesterol High (Investigations) | 1
Cardiac Troponin I Increased (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 1
White Blood Cell Decreased (Investigations) | 3
Alkaline Phosphatase Increased (Investigations) | 4
Alanine Aminotransferase Increased (Investigations) | 2
Activated Partial Thromboplastin Time Prolonged (Investigations) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seizure (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Nervous System Disorders - Other (Nervous system disorders) | 2
Ischemia Cerebrovascular (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hot Flashes (Vascular disorders) | 2
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03602586/Prot_SAP_000.pdf